CLINICAL TRIAL: NCT03471715
Title: Evaluation of Frequency of Root Fenestration and Dehiscence at Different Teeth Types in a Sample of Adult Egyptian Population Using Cone Beam Computed Tomography.
Brief Title: Frequency of Root Fenestration and Dehiscence in Adult Egyptian Population Using CBCT.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Prof. Nashwa Salah, professor of oral and axillofacia radiology faculty of dentistry, Cairo University
Other Study IDs: RAD 1:6:2
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Root Fenestation and Dehiscence
Keywords: frequency fenesration dehiscence cbct population

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
observational crosssectional study to evaluate the Frequency of Root Fenestration and Dehiscence at Different Teeth Types in a Sample of Adult Egyptian Population Using Cone Beam Computed Tomography.

DETAILED DESCRIPTION:
**Data Collection:

The following data of the current retrospective study will be collected from the recruited CBCT images:-

1. Demographic data:

   Age and Sex will be drawn from the patients' CBCT files.
2. Variables:

   Outcome: Frequency of root fenestration and dehiscence at different teeth types in adult Egyptian population sample using CBCT.

   Radiographic examination was done at the Oral and Maxillofacial Radiology Department, Faculty of Dentistry, Cairo University using CBCT machine, Planmeca Promax 3D Mid (Finland) .

   Root fenestration (RF) will be identified according to the definition of Davies et al. 19 and the American Association of Endodontists 20 as a tooth root protruding from a window-like opening or a defect in the alveolar bone without involvement of the alveolar margin. Three points should be emphasized in this definition. 1- A window-like opening or defect of the alveolar bone means that both the cortical bone and the cancellous bone are penetrated simultaneously, and the root either is in direct contact with the overlying mucosa or exposed to the oral environment. 2- The exposed root protrudes beyond the bone. 3- The exclusion of the alveolar margin emphasized to differentiate fenestration from dehiscence. While dehiscence will be identified as the crest of buccal and lingual bone that lies at least 4mm apical to the crest of interproximal bone.

   The identification and measurements of the alveolar bone level will be made on CBCT cross sectional images that are corrected to be with the long axis of each tooth under examination.

   All assessment will be done by two examiners to eliminate the inter-examiner error. All data regarding patient identification will be kept confidential.

   **Participants: Eligibility criteria
   1. Inclusion criteria:

      • CBCT scans of Adult Egyptian population with age range from 18 to 60 years old.

      • The CBCT scans should fully show both maxillary and mandibular teeth with the surrounding alveolar bone.

      • Permanent teeth with complete development of roots only are included.
      * CBCT scans for both partially and fully dentated people are included.
      * Lack of large pathological lesion.
      * Lack of fracture either in teeth or alveolar bone.
   2. Exclusion criteria:

      • CBCT scans of People younger than 18 or older than 60 years old.

      • CBCT scans showing only single jaw.

      • CBCT scans completely edentulous people.
      * Teeth with incomplete root development are excluded.
      * Teeth with unclear alveolar crest around it due to metallic artifacts from nearby restoration.
      * Presence of large pathological lesions.
      * Fractured teeth or alveolar process.

        * Sources:

      CBCT images will be obtained from patient's database at the Department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University.

      **Methods of selection: The sample will be selected by random manual means from database of Promax 3D Mid machine.

      **Bias: Investigators are going to be blinded about patients' age and gender prior to scans interpretation.
      * Blinding/Masking:

      After recruitment of images, a volunteering radiologist will perform coding of the images and clinical data. All investigators will be blinded of the data collected. The main investigator will evaluate the images twice with two weeks interval between the two reading sessions, while second investigator will evaluate it once. Inter-observational and intra-observational variability between the observers will be statistically evaluated.
      * Statistical Considerations:

      SAMPLE SIZE ESTIMATION This study is designed to determine the frequency of root fenestration and dehiscence at different teeth types in a sample of adult Egyptian population using CBCT. Based on previous study by Enhos et al (2012)13, Buyuk et al (2016) 21 and Gambarini et al (2017)15, the weighted average expected frequency of fenestration and dehiscence of the three studies are 7.0 % for fenestration and 4.8 % for dehiscence. A total sample size of 100 cases will be needed to provide a two-sided 95% confidence interval for a single proportion using the large sample normal approximation and will extend 5% from the observed proportion for an expected proportion of 0.07. Sample size estimation was performed by Epi info statistical package.

      STATISTICAL METHODS Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 23 (SPSS Inc., Chicago, IL). The estimation of the frequency of fenestration and dehiscence in a sample of the adult Egyptian population will be described as numbers and percentages. The 95% confidence intervals for all estimates will be calculated

ELIGIBILITY:
Inclusion Criteria:

* a- CBCT scans of Adult Egyptian population with age range from 18 to 60 years old.

  b- The CBCT scans should fully show both maxillary and mandibular teeth with the surrounding alveolar bone.

  c- Permanent teeth with complete development of roots only are included. d- CBCT scans for both partially and fully dentated people are included. e- Lack of large pathological lesion. f- Lack of fracture either in teeth or alveolar bone.

Exclusion Criteria:

1. CBCT scans of People younger than 18 or older than 60 years old.
2. CBCT scans showing only single jaw.
3. CBCT scans completely edentulous people.
4. Teeth with incomplete root development are excluded.
5. Teeth with unclear alveolar crest around it due to metallic artifacts from nearby restoration.
6. Presence of large pathological lesions.
7. Fractured teeth or alveolar process.

   -

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Frequency of Root Fenestration and Dehiscence at Different Teeth Types in a Sample of Adult Egyptian Population Using Cone Beam Computed Tomography. | 2016 2017 2018
  measuring device isCBCT machine, Planmeca Promax 3D Mid (Finland). unit is percentage %